CLINICAL TRIAL: NCT02672553
Title: A Randomized Comparison of the EDWARDS INTUITY Valve System anD commErcially Available Aortic Bioprostheses in Subjects uNdergoing surgiCal Aortic Valve Replacement Using Minimally InvaSive Techniques
Brief Title: EDWARDS INTUITY Valve System CADENCE-MIS Study
Acronym: CADENCE-MIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011-12
Record Dates: First submitted 2015-11-06; First posted 2016-02-03 (Estimated); Results first posted 2019-01-28 (Actual); Last update posted 2019-01-28 (Actual); Status verified 2018-08

CONDITIONS: Aortic Valve Disease; Aortic Stenosis
Keywords: Aortic Valve Replacement; Minimal Invasive Sternotomy
MeSH Terms: conditions — Aortic Valve Disease; Aortic Valve Stenosis | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- EDWARDS INTUITY (Active Comparator): EDWARDS INTUITY Valve System, Model 8300A
  Interventions: Device: EDWARDS INTUITY Valve System, Model 8300A
- Stented Aortic Bioprostheses (Active Comparator): Stented Aortic Bioprostheses
  Interventions: Device: Stented Aortic Bioprostheses

INTERVENTIONS:
Device: EDWARDS INTUITY Valve System, Model 8300A — To evaluate cardiac performance characteristics and adverse events rates associated with the EDWARDS INTUITY Valve in patients undergoing MIS-AVR.
  Other Names: aortic stenosis; stenosis-based insufficiency; aortic valve replacement
  Arms: EDWARDS INTUITY
Device: Stented Aortic Bioprostheses — In comparison to control valves available on the market undergoing FS-AVR
  Other Names: aortic stenosis; stenosis-based insufficiency; aortic valve replacement
  Arms: Stented Aortic Bioprostheses

SUMMARY:
The study purpose is to compare the EDWARDS INTUITY valve system in a minimal invasive surgical approach (MIS) with any commercially available aortic bioprosthesis in standard full sternotomy surgical approach.

DETAILED DESCRIPTION:
This is a randomized study to compare the cross-clamp time (XCT) and cardiopulmonary bypass time (CPBT) of the EDWARDS INTUITY valve system in a minimally invasive surgical approach (MIS) with any commercially available aortic bioprosthesis in standard full sternotomy surgical approach, in patients with logistic EuroScore < 20 undergoing elective isolated aortic valve replacement (AVR) surgery.

Additionally, the aim is to gather sufficient data to quantify the effect size of short term patient benefit outcomes previously identified from literature and to explore additional healthcare resource utilization endpoints.

ELIGIBILITY:
Inclusion:

1. adult male or female ≥18 years of age
2. symptomatic for aortic stenosis / mixed aortic stenosis and aortic insufficiency disease for which isolated surgical aortic valve replacement without concomitant procedures is planned
3. EuroSCORE <20
4. NYHA Class ≥II
5. Subject has signed and dated the investigation informed consent form prior to study specific procedures are performed
6. Subject is geographically stable and agrees to participate in follow-up assessments as specified in the protocol and informed consent

Exclusion (i.a.):

1. pure aortic insufficiency
2. previous cardiac surgery (involved FS or MIS approach)
3. congenital true bicuspid / unicuspid aortic valve
4. requires emergency surgery or has had emergency surgery for any reason

   ≤ 1 month before the intended treatment
5. LVEF <25%
6. active endocarditis ≤ 6 months before the intended treatment
7. acute MI ≤ 90 days before the intended treatment
8. had a stroke or transient ischemic attack within six months prior to scheduled aortic valve replacement surgery
9. oxygen or ventilator dependent
10. life expectancy < 12 months
11. substance abuser
12. Female subject is pregnant or lactating
13. documented leukopenia (WBC < 3.5x 103/μL), acute anemia (Hgb < 10.0 gm/dL or < 6.2 mmol/L), thrombocytopenia (platelet count < 100x 103/mL), or history of bleeding diathesis or coagulopathy
14. hemodynamic or respiratory instability requiring inotropic support, mechanical circulatory support, or mechanical ventilation within 30 days of procedure
15. documented echocardiographic evidence of intracardiac mass, thrombus or vegetation
16. renal insufficiency as determined by Serum creatinine ≥ 200 μmol/L (2.27 mg/dL) at screening or end-stage renal disease requiring chronic dialysis
17. documented hyperparathyroidism
18. currently participating in an investigational drug or device trial for which follow-up has not yet been completed
19. Minimally Invasive access to the heart is not possible due to anatomical constraints or any other pre-existing condition

Intra-operative Exclusion:

1. has calcium on the anterior mitral leaflet which cannot be removed
2. has extensive calcification of the aortic root
3. Annular deformation which may or may not be caused by too extensive decalcification of the aortic annulus
4. has left atrial thrombus
5. The position of the coronary ostia relative to the EDWARDS INTUITY Valve would result in obstruction of blood flow
6. hemodynamically unstable during the procedure requiring the procedure to be aborted prior to insertion of the study bioprosthesis and delivery system
7. Study device is not available in the correct size for the subject

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-05; Primary Completion 2015-03 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Borger, MD, Principal Investigator — Leipzig Heart Center
Locations (1):
- Leipzig Heart Center, Leipzig, Saxony, Germany

IPD SHARING:
Plan to Share IPD: No
As of this date no IPD plan has been formulated.

REFERENCES:
- [Result] Borger MA, Dohmen PM, Knosalla C, Hammerschmidt R, Merk DR, Richter M, Doenst T, Conradi L, Treede H, Moustafine V, Holzhey DM, Duhay F, Strauch J. Haemodynamic benefits of rapid deployment aortic valve replacement via a minimally invasive approach: 1-year results of a prospective multicentre randomized controlled trial. Eur J Cardiothorac Surg. 2016 Oct;50(4):713-720. doi: 10.1093/ejcts/ezw042. Epub 2016 Mar 2. PMID 26935407
- [Result] Borger MA, Moustafine V, Conradi L, Knosalla C, Richter M, Merk DR, Doenst T, Hammerschmidt R, Treede H, Dohmen P, Strauch JT. A randomized multicenter trial of minimally invasive rapid deployment versus conventional full sternotomy aortic valve replacement. Ann Thorac Surg. 2015 Jan;99(1):17-25. doi: 10.1016/j.athoracsur.2014.09.022. Epub 2014 Nov 20. PMID 25441065

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All eligible subjects recruited were randomized to each arm/group as 1:1 ratio at start.
Pre-assignment Details: Three (3) of the subjects randomized to the Edwards INTUITY group were converted to the control group and received a commercially available surgical aortic heart valve via MIS and therefore these three (3) subjects could not be accurately categorized into the MIS-AVR or FS-AVR category and were excluded from the as intended (AI) cohort.
Groups:
- Edwards INTUITY Surgical Aortic Heart Valve: Subject who received an Edwards INTUITY surgical aortic heart valve undergoing MIS-AVR
- Control Group - Commercial Surgical Aortic Heart Valve: Subject who received a commercially available surgical aortic heart valve undergoing FS-AVR
Period: Overall Study
Arm/Group | Edwards INTUITY Surgical Aortic Heart Valve | Control Group - Commercial Surgical Aortic Heart Valve
Started | 51 | 49
Intent To Treated (ITT) Randomized Arm (Intent to treat (ITT) is defined as the initial treatment assignment.) | 49 (Two (2) subjects randomized to Edwards INTUITY were intraoperative screen failures) | 48 (One (1) subject randomized to Control arm/group withdrew prior to study procedure)
As Treated (AT) Randomized Arm/Group | 46 | 51
As Intended (AI) Randomized Arm/Group (As intended (AI) excluded the three INTUITY subjects converted to control group from analysis.) | 46 | 48
Completed | 39 | 41
Not Completed | 12 | 8
Not completed — Death | 3 | 5
Not completed — Valve Explant | 1 | 0
Not completed — Conversion to Commercial Valve | 3 | 0
Not completed — Withdrawal by Subject | 3 | 3
Not completed — Intraoperative screen failure | 2 | 0

BASELINE CHARACTERISTICS:
Population: 3 of the subjs. randomized to the Edwards INTUITY group were converted to the control group and rec'd commercially available surgical aortic heart valves.From the overall,2 randomized to Edwards INTUITY &1 randomized to control group were screen failures prior to procedure & were excluded in the baseline analysis.Analysis is based on the AI cohort
Groups:
- Total: Total of all reporting groups
Arm/Group | Edwards INTUITY Surgical Aortic Heart Valve | Control Group - Commercial Surgical Aortic Heart Valve | Total
Number analyzed (Participants) | 46 | 48 | 94
Age, Continuous [Mean (Standard Deviation); unit: Years] | 73.0 (5.3) | 74.2 (5.0) | 73.61 (5.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 27 | 46
  Male | 27 | 21 | 48
Region of Enrollment [Count of Participants; unit: Participants]
  Europe | 46 | 48 | 94

OUTCOME MEASURES:

1. Primary Outcome: Median Subject Time Spent on Cardiopulmonary Cross Clamp
Description: Cardiopulmonary cross clamp time is the amount of time that the patient's aorta (blood vessel) is clamped by a surgical instrument used in cardiac surgery. This allows the normal blood flow to be sent to an artificial heart and lung machine to keep it at a constant temperature and oxygen level.
Time Frame: At time of surgery; an average of 1 hour
Population: The outcome is reported for subjects where data is available. Analysis is based on the AI cohort
Measure: Median (Full Range); unit: Minutes
Arm/Group | Edwards INTUITY Surgical Aortic Heart Valve | Control Group - Commercial Surgical Aortic Heart Valve
Number analyzed (Participants) | 46 | 48
Minutes | 35.0 [16.0 to 115.0] | 47.5 [32.0 to 123.0]
Statistical Analysis 1: Comparison: Edwards INTUITY Surgical Aortic Heart Valve vs Control Group - Commercial Surgical Aortic Heart Valve; Test type: Superiority; p < 0.0001, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = -12.5

2. Primary Outcome: Median Amount of Time Subject Spent on Cardiopulmonary Bypass
Description: Cardiopulmonary bypass time is the amount of time that the patient's blood circulates through an artificial heart and lung machine during cardiac surgery.
Time Frame: At time of surgery; an average of 1 hour
Population: The outcome is reported for subjects where data is available. Analysis is based on the AI cohort
Measure: Median (Full Range); unit: Minutes
Arm/Group | Edwards INTUITY Surgical Aortic Heart Valve | Control Group - Commercial Surgical Aortic Heart Valve
Number analyzed (Participants) | 46 | 48
Minutes | 58.5 [38.0 to 161.0] | 69.0 [39.0 to 170.0]
Statistical Analysis 1: Comparison: Edwards INTUITY Surgical Aortic Heart Valve vs Control Group - Commercial Surgical Aortic Heart Valve; Test type: Superiority; p = 0.2077, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = -10.5

3. Secondary Outcome: Number of Participants With Change From Baseline in New York Heart Association (NYHA) Class at 2 Years.
Description: The New York Heart Association (NYHA) functional classification system relates symptoms to everyday activities and the patient's quality of life.
  Class I. Patients with cardiac disease but without resulting limitation of physical activity.
  Class II. Patients with cardiac disease resulting in slight limitation of physical activity. They are comfortable at rest.
  Class III. Patients with cardiac disease resulting in marked limitation of physical activity. They are comfortable at rest.
  Class IV. Patients with cardiac disease resulting in inability to carry on any physical activity without discomfort. Symptoms of heart failure or the anginal syndrome may be present even at rest.
Time Frame: Baseline and 2 Years.
Population: The outcome is reported for subjects where data is available. Analysis is based on the ITT cohort
Measure: Count of Participants; unit: Participants
Arm/Group | Edwards INTUITY Surgical Aortic Heart Valve | Control Group - Commercial Surgical Aortic Heart Valve
Number analyzed (Participants) | 40 | 39
Participants
  Improved | 22 | 27
  Same | 17 | 11
  Worsened | 1 | 1

4. Secondary Outcome: Subject's Average Mean Gradients (mmHg) Measurements Over Time.
Description: Mean gradient is the average flow of blood through the aortic valve measured in millimeters of mercury. Gradients are evaluated by echocardiography over time. Mean gradient values depend on the size and type of valve.
Time Frame: Baseline, Discharge, 30 days, 3 Months, 1 Year
Population: The outcome is reported for subjects where data is available. Analysis is based on the AI cohort
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Edwards INTUITY Surgical Aortic Heart Valve | Control Group - Commercial Surgical Aortic Heart Valve
Number analyzed (Participants) | 46 | 48
mmHg
  Baseline: number analyzed (Participants) | 42 | 45
  Baseline | 44.0 (15.9) | 45.4 (20.0)
  Discharge: number analyzed (Participants) | 40 | 44
  Discharge | 10.3 (5.4) | 10.8 (3.4)
  30 days: number analyzed (Participants) | 33 | 37
  30 days | 8.8 (4.2) | 9.7 (3.9)
  3 months: number analyzed (Participants) | 39 | 40
  3 months | 9.1 (4.2) | 10.3 (4.8)
  1 year: number analyzed (Participants) | 40 | 40
  1 year | 9.1 (2.9) | 11.5 (4.3)

5. Secondary Outcome: Subject's Average Peak Gradients (mmHg) Measurements Over Time.
Description: Peak gradient is the maximum value measured of flow of blood through the aortic valve as measured in millimeters of mercury. Gradients are evaluated by echocardiography over time.
Time Frame: Baseline, Discharge, 30 days, 3 Months, 1 Year
Population: The outcome is reported for subjects where data is available. Analysis is based on the AI cohort
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Edwards INTUITY Surgical Aortic Heart Valve | Control Group - Commercial Surgical Aortic Heart Valve
Number analyzed (Participants) | 46 | 48
mmHg
  Baseline: number analyzed (Participants) | 42 | 45
  Baseline | 69.6 (23.7) | 75.4 (27.9)
  Discharge: number analyzed (Participants) | 40 | 44
  Discharge | 19.0 (9.5) | 21.0 (6.9)
  30 days: number analyzed (Participants) | 33 | 37
  30 days | 16.5 (7.8) | 17.8 (6.5)
  3 months: number analyzed (Participants) | 39 | 40
  3 months | 17.0 (7.6) | 18.9 (8.2)
  1 year: number analyzed (Participants) | 40 | 40
  1 year | 16.9 (5.3) | 21.9 (8.6)

6. Secondary Outcome: Subject's Effective Orifice Area (EOA) Measurement Over Time.
Description: Effective orifice area represents the cross-sectional area of the blood flow downstream of the aortic valve. Effective orifice area is evaluated by echocardiography over time.
Time Frame: Baseline, Discharge, 30 days, 3 Months, 1 Year
Population: The outcome is reported for subjects where data is available. Analysis is based on the AI cohort
Measure: Mean (Standard Deviation); unit: centimeters squared
Arm/Group | Edwards INTUITY Surgical Aortic Heart Valve | Control Group - Commercial Surgical Aortic Heart Valve
Number analyzed (Participants) | 46 | 48
centimeters squared
  Baseline: number analyzed (Participants) | 38 | 43
  Baseline | 0.7 (0.2) | 0.7 (0.2)
  Discharge: number analyzed (Participants) | 38 | 36
  Discharge | 1.9 (0.6) | 1.9 (0.7)
  30 days: number analyzed (Participants) | 30 | 31
  30 days | 1.9 (0.5) | 2.0 (0.7)
  3 months: number analyzed (Participants) | 36 | 39
  3 months | 1.9 (0.5) | 1.8 (0.6)
  1 year: number analyzed (Participants) | 27 | 29
  1 year | 1.9 (0.5) | 1.7 (0.4)

7. Secondary Outcome: Amount of Paravalvular Leak Over Time.
Description: Number of subjects who experienced a Paravalvular Leak shown over various time points.
  Paravalvular leak refers to blood flowing through a channel between the implanted artificial valve and the cardiac tissue as a result of inappropriate sealing.
  Paravalvular leak is evaluated by echocardiography over time. It is assessed on a scale from minimum of 0 to maximum of 4, where 0 = no leak, 1 = a trace leak, 2 = a mild leak, 3 = a moderate leak, and 4 = a severe leak.
  Higher numbers on the scale show a worsening outcome.
Time Frame: Discharge, 30 days, 3 month, 1 year
Population: The outcome is reported for subjects where data is available. Analysis is based on the AI cohort
Measure: Count of Participants; unit: Participants
Arm/Group | Edwards INTUITY Surgical Aortic Heart Valve | Control Group - Commercial Surgical Aortic Heart Valve
Number analyzed (Participants) | 46 | 48
Participants
  Discharge: number analyzed (Participants) | 41 | 43
  Discharge: 0 None | 30 | 33
  Discharge: +1 Trivial/Trace | 10 | 7
  Discharge: +2 Mild | 1 | 3
  Discharge: +3 Moderate | 0 | 0
  Discharge: +4 Severe | 0 | 0
  30 days: number analyzed (Participants) | 34 | 36
  30 days: 0 None | 27 | 24
  30 days: +1 Trivial/Trace | 6 | 11
  30 days: +2 Mild | 1 | 1
  30 days: +3 Moderate | 0 | 0
  30 days: +4 Severe | 0 | 0
  3 months: number analyzed (Participants) | 42 | 39
  3 months: 0 None | 26 | 27
  3 months: +1 Trivial/Trace | 13 | 9
  3 months: +2 Mild | 2 | 3
  3 months: +3 Moderate | 1 | 0
  3 months: +4 Severe | 0 | 0
  1 year: number analyzed (Participants) | 36 | 40
  1 year: 0 None | 23 | 34
  1 year: +1 Trivial/Trace | 9 | 6
  1 year: +2 Mild | 3 | 0
  1 year: +3 Moderate | 1 | 0
  1 year: +4 Severe | 0 | 0

8. Secondary Outcome: Conversion of Edwards INTUITY Surgical Aortic Valve to Control Surgical Aortic Heart Valves During Surgery.
Description: Subjects randomized to the Edwards INTUITY group that were converted to the control group and received commercially available surgical aortic heart valves during surgery.
Time Frame: Prior to Surgery
Population: Analysis is based on the ITT cohort
Measure: Count of Participants; unit: Participants
Arm/Group | Edwards INTUITY Surgical Aortic Heart Valve | Control Group - Commercial Surgical Aortic Heart Valve
Number analyzed (Participants) | 49 | 48
Participants | 3 | 0

9. Secondary Outcome: Subjects Who Required a Thoracic Resternotomy Over Time
Description: Number of Subjects who had a surgical opening of their chest after their initial aortic heart valve surgery shown over various time points.
Time Frame: 30 days, 3 Months, 1 Year, 2 Years.
Population: Cumulative number of subjects with an event by each time point Analysis is based on the AI cohort
Measure: Count of Participants; unit: Participants
Arm/Group | Edwards INTUITY Surgical Aortic Heart Valve | Control Group - Commercial Surgical Aortic Heart Valve
Number analyzed (Participants) | 46 | 48
Participants
  30 days | 6 | 5
  3 months | 6 | 5
  1 year | 7 | 5
  2 year | 7 | 5

10. Secondary Outcome: Subjects Who Received a Permanent Pacemaker Over Time.
Description: Number of Subjects who received a Permanent Pacemaker shown over various time points.
Time Frame: 30 days, 3 Months, 1 Year, 2 Years.
Population: Cumulative number of subjects with an event by each time point. Analysis is based on the AI cohort
Measure: Count of Participants; unit: Participants
Arm/Group | Edwards INTUITY Surgical Aortic Heart Valve | Control Group - Commercial Surgical Aortic Heart Valve
Number analyzed (Participants) | 46 | 48
Participants
  30 days | 2 | 1
  3 months | 2 | 1
  1 year | 2 | 1
  2 year | 3 | 2

11. Secondary Outcome: Subjects With a Paravalvular Leak > or Equal to 3+ and/or Requiring Intervention Over Time
Description: Number of subjects who experienced a Paravalvular Leak shown over various time points.
  Paravalvular leak refers to blood flowing through a channel between the implanted artificial valve and the cardiac tissue as a result of inappropriate sealing.
  Paravalvular leak is evaluated by echocardiography over time. It is assessed on a scale from 0 to 4, where 0 = no leak, 1 = a trace leak, 2 = a mild leak, 3 = a moderate leak, and 4 = a severe leak.
  Higher numbers on the scale show a worsening outcome.
Time Frame: 30 days, 3 Months, 1 Year, 2 Years.
Population: Cumulative number of subjects with an event by each time point. Analysis is based on the AI cohort
Measure: Count of Participants; unit: Participants
Arm/Group | Edwards INTUITY Surgical Aortic Heart Valve | Control Group - Commercial Surgical Aortic Heart Valve
Number analyzed (Participants) | 46 | 48
Participants
  30 days | 0 | 1
  3 months | 0 | 1
  1 year | 2 | 1
  2 year | 2 | 1

12. Secondary Outcome: Subjects Who Experienced Major Bleeding Over Time.
Description: Number of subjects who experienced Major Bleeding shown over various time points.
Time Frame: 30 days, 3 Months, 1 Year, 2 Years.
Population: Cumulative number of subjects with an event by each time point. Analysis is based on the AI cohort
Measure: Count of Participants; unit: Participants
Arm/Group | Edwards INTUITY Surgical Aortic Heart Valve | Control Group - Commercial Surgical Aortic Heart Valve
Number analyzed (Participants) | 46 | 48
Participants
  30 days | 8 | 4
  3 months | 8 | 5
  1 year | 8 | 5
  2 year | 8 | 5

13. Secondary Outcome: Subjects Who Experienced Respiratory Failure Over Time
Description: Number of subjects who experienced a Respiratory Failure shown over various time points. Respiratory failure happens when not enough oxygen passes from your lungs to your blood.
Time Frame: 30 days, 3 Months, 1 Year, 2 Years.
Population: Cumulative number of subjects with an event by each time point. Analysis is based on the AI cohort
Measure: Count of Participants; unit: Participants
Arm/Group | Edwards INTUITY Surgical Aortic Heart Valve | Control Group - Commercial Surgical Aortic Heart Valve
Number analyzed (Participants) | 46 | 48
Participants
  30 days | 2 | 0
  3 months | 2 | 0
  1 year | 2 | 2
  2 year | 2 | 2

14. Secondary Outcome: Subjects With a Cerebral Vascular Accident or Permanent Stroke Over Time
Description: Number of subjects who experienced a Cerebral Vascular Accident or Permanent Stroke shown over various time points.
Time Frame: 30 days, 3 Months, 1 Year, 2 Years.
Population: Cumulative number of subjects with an event by each time point. Analysis is based on the AI cohort
Measure: Count of Participants; unit: Participants
Arm/Group | Edwards INTUITY Surgical Aortic Heart Valve | Control Group - Commercial Surgical Aortic Heart Valve
Number analyzed (Participants) | 46 | 48
Participants
  30 days | 2 | 2
  3 months | 2 | 2
  1 year | 2 | 2
  2 year | 3 | 2

15. Secondary Outcome: Subjects With Renal Failure Over Time
Description: Number of subjects who experienced Renal (kidney) Failure shown over various time points.
Time Frame: 30 days, 3 Months, 1 Year, 2 Years.
Population: Cumulative number of subjects with an event by each time point. Analysis is based on the AI cohort
Measure: Count of Participants; unit: Participants
Arm/Group | Edwards INTUITY Surgical Aortic Heart Valve | Control Group - Commercial Surgical Aortic Heart Valve
Number analyzed (Participants) | 46 | 48
Participants
  30 days | 3 | 0
  3 months | 3 | 0
  1 year | 3 | 1
  2 year | 3 | 1

16. Secondary Outcome: Subjects With Endocarditis Over Time
Description: Number of subjects who experienced Endocarditis shown over various time points. Endocarditis is an infection of the endocardium, which is the inner lining of your heart chambers and heart valves.
Time Frame: 30 days, 3 Months, 1 Year, 2 Years.
Population: Cumulative number of subjects with an event by each time point. Analysis is based on the AI cohort
Measure: Count of Participants; unit: Participants
Arm/Group | Edwards INTUITY Surgical Aortic Heart Valve | Control Group - Commercial Surgical Aortic Heart Valve
Number analyzed (Participants) | 46 | 48
Participants
  30 days | 0 | 0
  3 months | 0 | 0
  1 year | 0 | 0
  2 year | 0 | 0

17. Secondary Outcome: Subjects With a Deep Sternal Would Infection Over Time
Description: Number of subjects who experienced a Deep Sternal Wound Infection shown over various time points.
Time Frame: 30 days, 3 Months, 1 Year, 2 Years.
Population: Cumulative number of subjects with an event by each time point. Analysis is based on the AI cohort
Measure: Count of Participants; unit: Participants
Arm/Group | Edwards INTUITY Surgical Aortic Heart Valve | Control Group - Commercial Surgical Aortic Heart Valve
Number analyzed (Participants) | 46 | 48
Participants
  30 days | 1 | 1
  3 months | 1 | 1
  1 year | 1 | 1
  2 year | 1 | 1

18. Secondary Outcome: Subjects With a Myocardial Infarction Over Time
Description: Number of subjects who experienced a Myocardial Infarction shown over various time points. A Myocardial infarction, commonly known as a heart attack, occurs when blood flow decreases or stops to a part of the heart, causing damage to the heart muscle.
Time Frame: 30 days, 3 Months, 1 Year, 2 Years.
Population: Cumulative number of subjects with an event by each time point. Analysis is based on the AI cohort
Measure: Count of Participants; unit: Participants
Arm/Group | Edwards INTUITY Surgical Aortic Heart Valve | Control Group - Commercial Surgical Aortic Heart Valve
Number analyzed (Participants) | 46 | 48
Participants
  30 days | 0 | 1
  3 months | 0 | 1
  1 year | 0 | 2
  2 year | 0 | 2

19. Secondary Outcome: Subjects With a Thromboembolism Over Time
Description: Number of subjects who experienced a Thromboembolism shown over various time points. A thromboembolism is an obstruction of a blood vessel by a blood clot that has become dislodged from another site in the circulation.
Time Frame: 30 days, 3 Months, 1 Year, 2 Years.
Population: Cumulative number of subjects with an event by each time point. Analysis is based on the AI cohort
Measure: Count of Participants; unit: Participants
Arm/Group | Edwards INTUITY Surgical Aortic Heart Valve | Control Group - Commercial Surgical Aortic Heart Valve
Number analyzed (Participants) | 46 | 48
Participants
  30 days | 3 | 3
  3 months | 3 | 3
  1 year | 4 | 4
  2 year | 5 | 4

20. Secondary Outcome: Subjects With a Cardiac Tamponade Over Time
Description: Number of subjects who experienced a Cardiac Tamponade shown over various time points. Cardiac tamponade is when fluid in the pericardium (the sac around the heart) builds up and results in compression (squeezing) of the heart.
Time Frame: 30 days, 3 Months, 1 Year, 2 Years.
Population: Cumulative number of subjects with an event by each time point. Analysis is based on the AI cohort
Measure: Count of Participants; unit: Participants
Arm/Group | Edwards INTUITY Surgical Aortic Heart Valve | Control Group - Commercial Surgical Aortic Heart Valve
Number analyzed (Participants) | 46 | 48
Participants
  30 days | 2 | 3
  3 months | 2 | 3
  1 year | 2 | 3
  2 year | 2 | 3

21. Secondary Outcome: Subjects With a Cardiac Reoperation for Any Reason Over Time
Description: Number of subjects who experienced a Cardiac reoperation for any reason shown over various time points.
Time Frame: 30 days, 3 Months, 1 Year, 2 Years.
Population: Cumulative number of subjects with an event by each time point. Analysis is based on the AI cohort
Measure: Count of Participants; unit: Participants
Arm/Group | Edwards INTUITY Surgical Aortic Heart Valve | Control Group - Commercial Surgical Aortic Heart Valve
Number analyzed (Participants) | 46 | 48
Participants
  30 days | 6 | 5
  3 months | 6 | 5
  1 year | 7 | 6
  2 year | 7 | 6

22. Secondary Outcome: Conversion of Subjects Undergoing Minimally Invasive Surgical Incision to Full Sternotomy for the Randomized to Edwards INTUITY Group During Surgery.
Description: Subjects Randomized to Edwards INTUITY Group's Surgical Aortic Valve undergoing Minimally Invasive Surgical incision being converted to a Full Sternotomy open procedure During Surgery.
Time Frame: Prior to Surgery
Population: Analysis is based on the ITT cohort
Measure: Count of Participants; unit: Participants
Arm/Group | Edwards INTUITY Surgical Aortic Heart Valve | Control Group - Commercial Surgical Aortic Heart Valve
Number analyzed (Participants) | 49 | 48
Participants | 0 | 0

23. Secondary Outcome: Subject's Average Score on the EQ-5D - Quality of Life Questionnaire Over Time
Description: The EuroQol-5 Dimension (EQ-5D) is a standardized questionnaire that asks subjects to rate themselves (no problems, some problems, extreme problems) on mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The scale is indexed and ranges from a minimum of 0.275 and a maximum of 1.000. A lower number indicates the participants experiences more problems and a higher number indicates the participants experiences fewer problems.
Time Frame: Baseline, 30 days, 3 Months, 1 Year
Population: The outcome is reported where data is available. Analysis is based on the ITT cohort
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Edwards INTUITY Surgical Aortic Heart Valve | Control Group - Commercial Surgical Aortic Heart Valve
Number analyzed (Participants) | 49 | 48
units on a scale
  Baseline: number analyzed (Participants) | 48 | 48
  Baseline | 0.900 (0.097) | 0.902 (0.087)
  30 day: number analyzed (Participants) | 38 | 39
  30 day | 0.862 (0.080) | 0.902 (0.094)
  3 month: number analyzed (Participants) | 44 | 42
  3 month | 0.908 (0.080) | 0.918 (0.077)
  1 year: number analyzed (Participants) | 42 | 42
  1 year | 0.922 (0.086) | 0.925 (0.086)

24. Secondary Outcome: Subject's Average Score SF-12 - Quality of Life Questionnaire Over Time
Description: Subject's Average Score at Baseline and at each follow-up interval until 2 year - SF-12.
  The Medical Outcomes Study Short-Form 12 (SF-12) - Physical Component Summary (PCS) and Mental Component Summary (MCS).
  The SF-12 questionnaire scale ranges from 100, which reflects the best health status to 0, which reflects the worse health status.
Time Frame: Baseline, 30 days, 3 Months, 1 Year
Population: The outcome is reported where data is available. Analysis is based on the ITT cohort
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Edwards INTUITY Surgical Aortic Heart Valve | Control Group - Commercial Surgical Aortic Heart Valve
Number analyzed (Participants) | 49 | 48
units on a scale
  PCS - Baseline: number analyzed (Participants) | 48 | 46
  PCS - Baseline | 42.39 (9.18) | 40.79 (9.96)
  PCS - 30 day: number analyzed (Participants) | 36 | 37
  PCS - 30 day | 36.16 (10.08) | 38.45 (7.86)
  PCS - 3 month: number analyzed (Participants) | 44 | 42
  PCS - 3 month | 41.42 (8.19) | 43.95 (7.88)
  PCS - 1 year: number analyzed (Participants) | 42 | 40
  PCS - 1 year | 43.84 (9.46) | 44.70 (8.39)
  MCS - Baseline: number analyzed (Participants) | 48 | 46
  MCS - Baseline | 48.02 (12.85) | 50.07 (11.80)
  MCS - 30 day: number analyzed (Participants) | 37 | 37
  MCS - 30 day | 48.06 (12.88) | 50.26 (11.78)
  MCS - 3 month: number analyzed (Participants) | 44 | 42
  MCS - 3 month | 49.87 (11.28) | 51.37 (9.76)
  MCS - 1 year: number analyzed (Participants) | 42 | 41
  MCS - 1 year | 51.08 (8.80) | 52.46 (8.58)

25. Secondary Outcome: Subject's Average Score on the KCCQ - Quality of Life Questionnaire Over Time
Description: The Kansas City Cardiomyopathy Questionnaire (KCCQ) is a 23-item, self-administered instrument that quantifies physical function, symptoms (frequency, severity and recent change), social function, self-efficacy and knowledge, and quality of life. Scores range from 0-100, in which higher scores reflect better health status. Subjects took this questionnaire at Baseline, 30 days, 3 Months,and 1 Year.
Time Frame: Baseline, 30 days, 3 Months, 1 Year
Population: The outcome is reported where data is available. Analysis is based on the ITT cohort
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Edwards INTUITY Surgical Aortic Heart Valve | Control Group - Commercial Surgical Aortic Heart Valve
Number analyzed (Participants) | 49 | 48
units on a scale
  Baseline: number analyzed (Participants) | 49 | 46
  Baseline | 58.37 (24.79) | 61.33 (24.20)
  30 day: number analyzed (Participants) | 38 | 39
  30 day | 57.81 (23.64) | 64.33 (24.90)
  3 month: number analyzed (Participants) | 44 | 42
  3 month | 69.32 (23.58) | 76.35 (19.91)
  1 year: number analyzed (Participants) | 42 | 41
  1 year | 73.85 (21.25) | 78.11 (21.05)

26. Secondary Outcome: Health Care Utilization
Description: The average amount of time the subjects spent in the intensive care unit, the intermediate care length of stay, and the average total length of hospital stay after their heart valve replacement procedure.
Time Frame: Day of surgical procedure through discharge from the hospital, an average of 1.5 weeks
Population: This outcome is reported for subjects where data is available. Analysis is based on the ITT cohort
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Edwards INTUITY Surgical Aortic Heart Valve | Control Group - Commercial Surgical Aortic Heart Valve
Number analyzed (Participants) | 49 | 48
Days
  Length of stay | 10.9 (7.0) | 11.5 (9.2)
  ICU Length of stay: number analyzed (Participants) | 47 | 48
  ICU Length of stay | 2.6 (5.4) | 1.6 (1.5)
  Intermediate Care Length of stay: number analyzed (Participants) | 47 | 48
  Intermediate Care Length of stay | 1.3 (1.7) | 0.9 (1.3)

27. Secondary Outcome: Subject's Effective Orifice Area Index (EOAI) Measurement Over Time.
Description: Effective orifice area index represents the minimal cross-sectional area of the blood flow downstream of the aortic valve divided by the person's body surface area. Effective orifice area index is evaluated by echocardiography over time.
Time Frame: Baseline, Discharge, 30 days, 3 Months, 1 Year
Population: The outcome is reported for subjects where data is available. Analysis is based on the AI cohort
Measure: Mean (Standard Deviation); unit: centimeters squared/meters squared
Arm/Group | Edwards INTUITY Surgical Aortic Heart Valve | Control Group - Commercial Surgical Aortic Heart Valve
Number analyzed (Participants) | 46 | 48
centimeters squared/meters squared
  Baseline: number analyzed (Participants) | 38 | 43
  Baseline | 0.4 (0.1) | 0.4 (0.1)
  Discharge: number analyzed (Participants) | 38 | 35
  Discharge | 0.9 (0.3) | 1.0 (0.4)
  30 days: number analyzed (Participants) | 27 | 31
  30 days | 1.0 (0.3) | 1.1 (0.3)
  3 months: number analyzed (Participants) | 36 | 39
  3 months | 1.0 (0.2) | 1.0 (0.3)
  1 year: number analyzed (Participants) | 27 | 29
  1 year | 1.0 (0.3) | 0.9 (0.2)

28. Secondary Outcome: Amount of Aortic Valvular Regurgitation Over Time.
Description: Aortic valvular regurgitation occurs when the aortic valve in the heart does not close tightly allowing some of the blood that was pumped out of the heart to leak back into it. Aortic valvular regurgitation is evaluated by echocardiography over time. It is assessed on a scale from 0 to 4, where 0 represents no regurgitation and 4 represents severe regurgitation.
  Higher numbers on the scale show a worsening outcome.
Time Frame: Discharge, 30 days, 3 month, 1 year
Population: The outcome is reported for subjects where data is available. Analysis is based on the AI cohort
Measure: Count of Participants; unit: Participants
Arm/Group | Edwards INTUITY Surgical Aortic Heart Valve | Control Group - Commercial Surgical Aortic Heart Valve
Number analyzed (Participants) | 46 | 48
Participants
  Discharge: number analyzed (Participants) | 40 | 44
  Discharge: 0 None | 29 | 29
  Discharge: +1 Trivial/Trace | 10 | 13
  Discharge: +2 Mild | 1 | 2
  Discharge: +3 Moderate | 0 | 0
  Discharge: +4 Severe | 0 | 0
  30 days: number analyzed (Participants) | 35 | 38
  30 days: 0 None | 25 | 29
  30 days: +1 Trivial/Trace | 10 | 6
  30 days: +2 Mild | 0 | 3
  30 days: +3 Moderate | 0 | 0
  30 days: +4 Severe | 0 | 0
  3 months: number analyzed (Participants) | 43 | 40
  3 months: 0 None | 27 | 25
  3 months: +1 Trivial/Trace | 13 | 13
  3 months: +2 Mild | 2 | 2
  3 months: +3 Moderate | 1 | 0
  3 months: +4 Severe | 0 | 0
  1 year: number analyzed (Participants) | 40 | 40
  1 year: 0 None | 25 | 28
  1 year: +1 Trivial/Trace | 10 | 11
  1 year: +2 Mild | 5 | 1
  1 year: +3 Moderate | 0 | 0
  1 year: +4 Severe | 0 | 0

ADVERSE EVENTS:
Time Frame: Events occurring from baseline through two (2) years post implant
Description: Adverse event table is reported using ITT cohort
Arm/Group | Edwards INTUITY Surgical Aortic Heart Valve | Control Group - Commercial Surgical Aortic Heart Valve
All-Cause Mortality (participants affected / at risk) | 4/49 | 4/48
Serious Adverse Events (participants affected / at risk) | 31/49 | 27/48
Other Adverse Events (participants affected / at risk) | 27/49 | 30/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Edwards INTUITY Surgical Aortic Heart Valve (N=49) | Control Group - Commercial Surgical Aortic Heart Valve (N=48)
BLEEDING - CARDIOVASCULAR - MAJOR (Blood and lymphatic system disorders) | 4 | 1
BLEEDING - GASTROINTESTINAL UPPER -MAJOR (Blood and lymphatic system disorders) | 1 | 0
BLEEDING - NEUROLOGICAL - MAJOR (E.G. CVA) (Blood and lymphatic system disorders) | 1 | 1
BLEEDING - PERIPHERAL VASCULAR - MINOR (E.G. NOSEBLEEDS; HEMATOMAS) (Blood and lymphatic system disorders) | 1 | 0
THROMBOEMBOLIC EVENT - OTHER - CENTRAL - NO PARESIS (Cardiac disorders) | 0 | 1
THROMBOEMBOLIC EVENT - STROKE (Cardiac disorders) | 2 | 1
THROMBOEMBOLIC EVENT - TRANSIENT ISCHEMIC ATTACK (TIA) (Cardiac disorders) | 2 | 1
ARRHYTHMIA - PAROXYSMAL ATRIAL FIBRILLATION (PAF) (Cardiac disorders) | 4 | 4
ARRHYTHMIA - AV BLOCK - 3RD DEGREE (Cardiac disorders) | 2 | 2
ARRHYTHMIA - BRADYCARDIA (Cardiac disorders) | 0 | 1
ARRHYTHMIA - PERSISTANT ATRIAL FIBRILLATION (Cardiac disorders) | 1 | 1
ARRHYTHMIA - SUPRAVENTRICULAR TACHYCARDIA (SVT) (Cardiac disorders) | 0 | 1
ARRHYTHMIA - TACHYCARDIA - NON-VENTRICULAR (Cardiac disorders) | 0 | 1
ARRHYTHMIA - TACHYCARDIA - VENTRICULAR (Cardiac disorders) | 1 | 0
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 | 2
PERICARDIAL EFFUSION - MAJOR (Cardiac disorders) | 3 | 0
PERICARDIAL TAMPONADE - MAJOR (Cardiac disorders) | 2 | 3
CARDIAC DECOMPENSATION (Cardiac disorders) | 1 | 2
CARDIAC ARREST (Cardiac disorders) | 1 | 0
CARDIOVASCULAR - OTHER (Cardiac disorders) | 2 | 1
CARDIOGENIC SHOCK (Cardiac disorders) | 1 | 0
ENDOCARDITIS (Cardiac disorders) | 0 | 1
PERICARDITIS (Cardiac disorders) | 0 | 1
REGURGITATION - MITRAL-INDETERMINATE-+4 (Cardiac disorders) | 0 | 1
NSD - PARAVALVULAR LEAK - +4 (General disorders) | 1 | 0
NSD - PARAVALVULAR LEAK WITH HEMOLYSIS (General disorders) | 1 | 0
BILIARY (GALLBLADDER) (Gastrointestinal disorders) | 1 | 2
GASTROINTESTINAL - OTHER (Gastrointestinal disorders) | 3 | 2
GASTROINTESTINAL - INFECTION (Gastrointestinal disorders) | 1 | 0
GENITOURINARY - OTHER (Renal and urinary disorders) | 3 | 0
RENAL DYSFUNCTION (Renal and urinary disorders) | 0 | 1
RENAL FAILURE - ACUTE (Renal and urinary disorders) | 2 | 1
RENAL - OTHER (Renal and urinary disorders) | 1 | 0
URINARY TRACT INFECTION (UTI) (Renal and urinary disorders) | 1 | 0
MUSCULAR SKELETAL / DERMATOLOGIC - OTHER (Musculoskeletal and connective tissue disorders) | 2 | 6
STERNAL WOUND/THORACIC INFECTION (Musculoskeletal and connective tissue disorders) | 2 | 2
INFECTION /INFLAMMATION - OTHER (Musculoskeletal and connective tissue disorders) | 1 | 0
CANCER - NEWLY DIAGNOSED (General disorders) | 2 | 1
NONSPECIFIC, UNKNOWN, OR OTHER BODY SYSTEM - OTHER COMPLICATION (General disorders) | 2 | 3
ALLERGIC REACTION - MEDICATION RELATED (General disorders) | 0 | 1
MULTI-SYSTEM ORGAN FAILURE (General disorders) | 1 | 0
VASCULAR - OTHER (Vascular disorders) | 2 | 0
TRANSIENT PSYCHOTIC SYNDROME (Psychiatric disorders) | 1 | 1
PLEURAL EFFUSION - BILATERAL (Respiratory, thoracic and mediastinal disorders) | 5 | 3
RESPIRATORY INFECTION - PNEUMONIA (Respiratory, thoracic and mediastinal disorders) | 3 | 2
RESPIRATORY FAILURE -PNEUMONIA (Respiratory, thoracic and mediastinal disorders) | 1 | 2
PLEURAL EFFUSION - LEFT (Respiratory, thoracic and mediastinal disorders) | 2 | 0
RESPIRATORY FAILURE -COPD (Respiratory, thoracic and mediastinal disorders) | 1 | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Edwards INTUITY Surgical Aortic Heart Valve (N=49) | Control Group - Commercial Surgical Aortic Heart Valve (N=48)
ARRHYTHMIA - PAROXYSMAL ATRIAL FIBRILLATION (PAF) (Cardiac disorders) | 4 | 6
ARRHYTHMIA - PERMANENT ATRIAL FIBRILLATION (Cardiac disorders) | 0 | 3
PERICARDIAL EFFUSION - MINOR (Cardiac disorders) | 3 | 5
GASTROINTESTINAL - OTHER (Gastrointestinal disorders) | 1 | 3
MUSCULAR SKELETAL / DERMATOLOGIC - OTHER (Musculoskeletal and connective tissue disorders) | 5 | 5
PLEURAL EFFUSION - BILATERAL (Respiratory, thoracic and mediastinal disorders) | 2 | 3
ANEMIA - NON-BLEEDING RELATED (Blood and lymphatic system disorders) | 1 | 2
ANEMIA - BLEEDING RELATED - MINOR (Blood and lymphatic system disorders) | 0 | 1
BLEEDING - GASTROINTESTINAL LOWER -MINOR (Blood and lymphatic system disorders) | 1 | 0
BLEEDING - PULMONARY/RESPIRATORY MINOR (E.G. HEMOTHORAX) (Blood and lymphatic system disorders) | 1 | 0
BLOOD/ LYMPHATIC - OTHER (Blood and lymphatic system disorders) | 1 | 0
THROMBOEMBOLIC EVENT - TRANSIENT ISCHEMIC ATTACK (TIA) (Cardiac disorders) | 0 | 1
ARRHYTHMIA - ATRIAL FLUTTER (Cardiac disorders) | 1 | 0
ARRHYTHMIA - AV BLOCK - 1ST DEGREE (Cardiac disorders) | 1 | 1
ARRHYTHMIA - AV BLOCK - 2ND DEGREE (Cardiac disorders) | 0 | 1
ARRHYTHMIA - AV BLOCK - 3RD DEGREE (Cardiac disorders) | 0 | 1
ARRHYTHMIA - BRADYCARDIA (Cardiac disorders) | 1 | 0
ARRHYTHMIA - PAROXYSMAL ATRIAL TACHYCARDIA (PAT) (Cardiac disorders) | 1 | 0
ARRHYTHMIA - SUPRAVENTRICULAR TACHYCARDIA (SVT) (Cardiac disorders) | 1 | 1
ARRHYTHMIA - PERSISTANT ATRIAL FIBRILLATION (Cardiac disorders) | 0 | 1
ARRHYTHMIA - TACHYCARDIA - NON-VENTRICULAR (Cardiac disorders) | 1 | 0
CARDIOVASCULAR - OTHER (Cardiac disorders) | 1 | 1
NSD - PARAVALVULAR LEAK - +1 (General disorders) | 1 | 0
GASTROINTESTINAL - INFECTION (Gastrointestinal disorders) | 1 | 1
RENAL FAILURE - ACUTE (Renal and urinary disorders) | 1 | 2
GENITOURINARY - OTHER (Renal and urinary disorders) | 0 | 1
URINARY TRACT INFECTION (UTI) (Renal and urinary disorders) | 2 | 1
WOUND INFECTION - OTHER (Musculoskeletal and connective tissue disorders) | 0 | 1
INFECTION /INFLAMMATION - OTHER (Musculoskeletal and connective tissue disorders) | 1 | 0
NONSPECIFIC, UNKNOWN, OR OTHER BODY SYSTEM - OTHER COMPLICATION (General disorders) | 1 | 2
TRANSIENT PSYCHOTIC SYNDROME (Psychiatric disorders) | 2 | 2
PLEURAL EFFUSION - LEFT (Respiratory, thoracic and mediastinal disorders) | 2 | 1
PLEURAL EFFUSION - RIGHT (Respiratory, thoracic and mediastinal disorders) | 2 | 1
ATELECTASIS (Respiratory, thoracic and mediastinal disorders) | 1 | 1
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 2 | 0
PULMONARY/RESPIRATORY - OTHER (Respiratory, thoracic and mediastinal disorders) | 1 | 0
RESPIRATORY FAILURE -COPD (Respiratory, thoracic and mediastinal disorders) | 1 | 0
RESPIRATORY INFECTION - PNEUMONIA (Respiratory, thoracic and mediastinal disorders) | 1 | 1
RESPIRATORY FAILURE -OTHER (Respiratory, thoracic and mediastinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI can't publish/present on overall study results not yet published but may publish his own data subject to EW review prior to submission/presentation, but data analyses of site-specific results can occur only in intervals as specified in the CTA. Publication/presentation of the PI's site-specific results of devices which haven't been market released and which still may be undergoing development, shall not include claims of device safety/effectiveness and will require the review/approval of EW.